CLINICAL TRIAL: NCT00550888
Title: Comparison of Uterine Exteriorization Versus in Situ Repair at Cesarean Section: a Randomized Clinical Trial
Acronym: EXT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: IMIP1234
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2007-08

CONDITIONS: Cesarean Section
Keywords: uterus; abdominal delivery; suture techniques
MeSH Terms: interventions — Suture Techniques

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Procedure: suture techniques

SUMMARY:
There is no difference between extra-abdominal or in situ suture of the uterus in cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* indication of cesarean section
* gestational age > 24 weeks

Exclusion Criteria:

* two or more cesarean sections
* chorioamnionitis
* hemorrhagic complications
* unable to consent
* previous abdominal surgery

Ages: 13 Years to 44 Years | Sex: Female
Age Groups: Child, Adult
Dates: Start 2005-08; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
endometritis | within the first 30 days after surgery

SECONDARY OUTCOMES:
nausea and vomiting during surgery, mean operative time, estimated intraoperative blood loss, number of surgical sutures for uterine repair, pain postoperative, number of postoperative analgesic doses, surgical site infection | from surgery to 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Eronildo F Silva, Study Director — IMIP
Locations (1):
- IMIP Prof. Fernando Figueira, Recife, Pernambuco, Brazil

REFERENCES:
- [Derived] Coutinho IC, Ramos de Amorim MM, Katz L, Bandeira de Ferraz AA. Uterine exteriorization compared with in situ repair at cesarean delivery: a randomized controlled trial. Obstet Gynecol. 2008 Mar;111(3):639-47. doi: 10.1097/AOG.0b013e31816521e2. PMID 18310366